CLINICAL TRIAL: NCT02740491
Title: Evaluation of the Implementation of a "Remission" Consultation in the Management of Patients Treated for Localized Breast Cancer
Brief Title: Implementation of a "Remission" Consultation in the Management of Patients Treated for Localized Breast Cancer
Acronym: REVIS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2016/LD-01
Record Dates: First submitted 2016-04-07; First posted 2016-04-15 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- The study population: The study population consists of adult patients diagnosed with localized breast cancer who have completed adjuvant treatment (chemotherapy, radiotherapy) and who are cared for in the Medical Oncology department of the Nîmes University Hospital.
  Interventions: Other: Remission Consultation

INTERVENTIONS:
Other: Remission Consultation — At the end of adjuvant treatment (adjuvant chemotherapy and / or radiotherapy), the patient is seen by a referent oncologist and included in the study. A "Remission" consultation with a psychotherapist is then proposed and its purpose explained to the patient. The patient agrees or refuses take advantage of the "Remission" consultation; in case of refusal, the reasons are documented and further information is provided, thus giving the opportunity for the patient to benefit from further psychological counseling if desired.
  If approval is given, the patient will be scheduled for the "Remission" consultation (duration 1 hour) . The latter includes a first phase evaluating the mental state of the patient, and then a proposal of individualized care if necessary and according to several methods, depending on the choice of the patient.

SUMMARY:
The main objective of this study is to describe the evolution in quality of life (QLQ-C30) for patients receiving breast cancer care at 3, 6 and 12 months after a "remission" consultation.

DETAILED DESCRIPTION:
The secondary objectives of this study are:

A. to describe changes in body image (Image Body Scale Version F) at 3, 6 and 12 months after a "remission" consultation.

B. to describe changes in psychological distress (visual analog scale) at 3, 6 and 12 months after a "remission" consultation.

C. to assess the time of resumption of work (date of last chemotherapy - date of the actual resumption of work) after a "remission" consultation.

D. to evaluate the acceptance rate for the "remission" consultation.

E. to describe the modes of the observed management, their distribution and the characteristics of the patients according to different monitoring arrangements.

ELIGIBILITY:
Inclusion Criteria:

* The patient is receiving care for localized breast cancer and finished her adjuvant treatment (chemotherapy, radiotherapy)
* The patient has completed his/her adjuvant therapy in the last 6 months (chemotherapy, radiotherapy).

Exclusion Criteria:

* The patient is participating in another study
* The patient is under judicial protection
* It is impossible to correctly inform the patient
* The patient has a metastatic form of the disease at diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients diagnosed with localized breast cancer who have completed adjuvant treatment (chemotherapy, radiotherapy) and who are cared for in the Medical Oncology department of the Nîmes University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2019-10-24 (Actual)

PRIMARY OUTCOMES:
The EORTC QLQ-C30 questionnaire | Day 0
The EORTC QLQ-C30 questionnaire | Month 3
The EORTC QLQ-C30 questionnaire | Month 6
The EORTC QLQ-C30 questionnaire | Month 12

SECONDARY OUTCOMES:
Body Image Scale | Day 0
Body Image Scale | Month 3
Body Image Scale | Month 6
Body Image Scale | Month 12
Psychological distress (visual analog scale) | Day 0
Psychological distress (visual analog scale) | Month 3
Psychological distress (visual analog scale) | Month 6
Psychological distress (visual analog scale) | Month 12
Work recovery time (date of last chemotherapy - date of the actual resumption of work) | Month 3
Work recovery time (date of last chemotherapy - date of the actual resumption of work) | Month 6
Work recovery time (date of last chemotherapy - date of the actual resumption of work) | Month 12
Acceptance of remission consultation (yes/no) | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Luc Duwig, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] Alonso S, Kabani S, Fabbro-Peray P, Houede N, Duwig L. A feasibility study of scheduling a remission consultation in the management of patients treated for localized breast cancer. BMC Psychol. 2025 Sep 29;13(1):1087. doi: 10.1186/s40359-025-03393-6. PMID 41024190